CLINICAL TRIAL: NCT05842941
Title: HEALEY ALS Platform Trial - Regimen G DNL343
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518G
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Regimen Specific Appendix; Lou Gehrig's Disease; DNL343; Denali Therapeutics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DNL343 (Experimental)
  Interventions: Drug: DNL343
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: DNL343 — DNL343 is administered orally once daily per day for 24 weeks.
  Arms: DNL343
Drug: Matching Placebo — Matching placebo is administered orally once daily per day for 24 weeks.
  Arms: Matching Placebo

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

Regimen G will evaluate the safety and efficacy of a single study drug, DNL343, in participants with ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The HEALEY ALS Platform Trial Master Protocol is registered as NCT04297683. Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

If a participant is randomized to Regimen G DNL343, the participant will complete a screening visit to assess additional Regimen G eligibility criteria. Once Regimen G eligibility criteria are confirmed, participants will complete a baseline assessment and be randomized in a 3:1 ratio to either active DNL343 or matching placebo.

Regimen G will enroll by invitation, as participants may not choose to enroll in Regimen G. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen G.

For a list of enrolling sites, please see the HEALEY ALS Platform Trial Master Protocol under NCT04297683.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT NCT04297683).

Exclusion Criteria:

* The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT NCT04297683).

  1. Diagnosis of epilepsy or seizure within 6 months of randomization
  2. Hypersensitivity to DNL343 or any of the excipients contained within the DNL343 drug product
  3. The concomitant use of prescription or over-the-counter (OTC) medications that are inducers of certain cytochrome P450 enzymes, substrates of certain cytochrome P450 enzymes, or substrates of certain drug transporters.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Healey Center for ALS at Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DNL343: DNL343 is administered orally once a day for 24 weeks.
- Matching Placebo: Matching Placebo is administered orally once a day for 24 weeks.
Period: Overall Study
Arm/Group | DNL343 | Matching Placebo
Started | 186 | 63
Completed | 156 | 55
Not Completed | 30 | 8

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes only placebo participants from the Regimen G Efficacy Regimen Only (ERO) sample; shared placebo participants from other regimens are not included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | DNL343 | Matching Placebo | Total
Number analyzed (Participants) | 186 | 63 | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (11.55) | 57.3 (11.92) | 58.94 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 13 | 95
  Male | 104 | 50 | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 175 | 61 | 236
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 5 | 20
  Not Hispanic or Latino | 169 | 57 | 226
  Unknown or Not Reported | 2 | 1 | 3
ALS Diagnosis from R El Escorial Criteria [Count of Participants; unit: Participants] — The El Escorial Criteria are a set of guidelines used to diagnose ALS based on clinical signs of upper motor neuron and lower motor neuron dysfunction.
  Participants
    Clinically Possible ALS | 20 | 5 | 25
    Clinically Probable ALS - Laboratory Supported | 36 | 10 | 46
    Clinically Probable ALS | 62 | 26 | 88
    Clinically Definite ALS | 68 | 22 | 90
ALS Onset Location [Count of Participants; unit: Participants]
  Axial | 1 | 0 | 1
  Bulbar | 29 | 6 | 35
  Generalized | 0 | 0 | 0
  Limb | 155 | 56 | 211
  Multiple | 1 | 1 | 2
  Respiratory | 0 | 0 | 0
Time Since Symptom Onset at Baseline [Mean (Standard Deviation); unit: Months] | 19.7 (8.05) | 21.0 (7.91) | 20.1 (8.02)
Delay in ALS Symptom Onset and Diagnosis [Mean (Standard Deviation); unit: Months] | 10.3 (6.24) | 10.8 (5.68) | 10.4 (6.10)
Baseline Edaravone Use [Count of Participants; unit: Participants]
  Yes | 115 | 40 | 155
  No | 71 | 23 | 94
Baseline Riluzole Use [Count of Participants; unit: Participants]
  Yes | 161 | 54 | 215
  No | 25 | 9 | 34
Baseline Relyvrio Use [Count of Participants; unit: Participants]
  Yes | 102 | 35 | 137
  No | 84 | 28 | 112
ALSFRS-R Total Score [Mean (Standard Deviation); unit: Points] — The ALS Functional Rating Score-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Participants with higher scores have more physical function.
  Points | 36.0 (6.31) | 36.0 (5.91) | 36.0 (6.20)
Pre-Baseline Decline in ALSFRS-R [Mean (Standard Deviation); unit: Points per Month] — The decline score is 48-Baseline is divided by the number of months between onset of weakness due to ALS and the date of Baseline. A higher number indicates greater decline.
  Points per Month | 0.69 (0.441) | 0.70 (0.609) | 0.69 (0.49)
SVC [Mean (Standard Deviation); unit: Percent Predicted] — Slow vital capacity is an assessment of breathing function. The total amount of air that can be exhaled is measured. A higher slow vital capacity indicates better breathing function. Population: Number analyzed in row differs from overall number due to missing data.
  Percent Predicted
    number analyzed (Participants) | 185 | 63 | 248
    (all) | 85.0 (18.91) | 83.6 (15.05) | 84.7 (17.99)
King Stage [Count of Participants; unit: Participants] — The King's ALS Clinical Staging System is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction. Level 4a indicates nutritional failure and level 4b indicates respiratory failure. Higher scores indicate a worse disease state.
  Participants
    1 Region with Neuromuscular Dysfunction | 35 | 14 | 49
    2 Region with Neuromuscular Dysfunction | 47 | 9 | 56
    3 Region with Neuromuscular Dysfunction | 52 | 18 | 70
    4a/b Nutritional/Respiratory Failure | 52 | 22 | 74
Weight [Mean (Standard Deviation); unit: Kg] | 78.5 (16.49) | 82.4 (14.44) | 79.5 (16.06)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.54) | 26.3 (4.05) | 26.3 (4.42)
Serum Creatinine Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Number analyzed in row differs from overall number due to missing data.
  mg/dL
    number analyzed (Participants) | 185 | 62 | 247
    (all) | 0.7 (0.20) | 0.7 (0.16) | 0.7 (0.19)
Serum NfL Concentration [Median (Inter-Quartile Range); unit: ng/L] — Population: Number analyzed in row differs from overall number due to missing data.
  ng/L
    number analyzed (Participants) | 184 | 62 | 246
    (all) | 61.8 [42.1 to 90.0] | 50.7 [33.4 to 75.5] | 59.0 [40.3 to 87.1]

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Assessed by the ALSFRS-R-Slope
Description: Change in disease severity as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) total score using a Bayesian repeated measures model that accounts for loss to follow-up due to mortality. Each of 12 questions assessing distinct functional ability is scored from 4(normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Participants with higher scores have more physical function. Note that only participants who survived to their Week 24 visit contribute to the estimate.
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Efficacy Concurrent-controls Set (ECC), which included concurrent shared placebos from other regimens if randomized within 180 days of the first and last randomization for the applicable regimen, excluding any shared placebos also include in the focal regimen, as pre-specified in the Regimen Statistical Analysis Plan. Regimen F (NCT#05740813) and Regimen G (NCT#05842941) contributed placebo participants into the shared placebo cohort used for analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Percent change | -0.88 (0.062) | -0.84 (0.081)
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter model — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. (DNL343 slowed progression) was 0.3286. NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 1.06, 95% CI 2-sided [0.840 to 1.351], Standard Deviation 0.129 — DDR <1 imply slowing of disease progression by DNL343 relative to placebo. Note: reported "Confidence Interval" is actually a Bayesian credible interval; The DRR parameter for active treatment represents the relative change to the rate of decline of ALSFRS-R and the rate of mortality of treated participant relative to a placebo participant. The estimated DRR can also be interpreted as the average rate of decline in function and mortality. The model incorporates participant-level random effects in the baseline value of the ALSFRS-R (intercept) and in the rate of progression (slope); covariate effects to account for covariate-explainable differences in rates of progression based on participant-specific baseline covariates; regimen-specific differences in baseline values, rates of progression and measurement error. Covariates include baseline TRICALS score, log-transformed baseline serum NfL, riluzole, edaravone, and Relyvrio use at the time of baseline as indicated in concomitant medication logs

2. Secondary Outcome: ALSFRS-R Total Score
Description: Change in ALSFRS-R total score over time. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Participants with higher scores have more physical function.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Points
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Points | -5.759 (0.3810) | -5.726 (0.4325)
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.9562, Mixed Models Analysis; Covariates: baseline (BL) of use edaravone, riluzole, & Relyvrio, BL log NfL, SVC and TRICALS score and interaction with visit; Mean Difference (Net) = -0.033, 95% CI 2-sided [-1.203 to 1.137], Standard Error of Mean 0.5949; DNL343 24-week change from baseline relative to placebo 24-week change from baseline. The model include fixed terms for regimen, visit, treatment group, treatment group × visit interaction, baseline score and baseline score x visit interaction, baseline TRICALs risk score and baseline TRICALS risk score × visit interaction, baseline riluzole use and baseline riluzole use × visit interaction, baseline edaravone use and baseline edaravone use × visit interaction, baseline Relyvrio use and baseline Relyvrio × visit interaction, and baseline log-transformed serum NfL level and baseline log-transformed serum NfL level × visit interaction

3. Secondary Outcome: Combined Assessment of Function and Survival (CAFS)
Description: Combined assessment of function and survival (CAFS) ranks participants' clinical outcomes based on survival time and change in the functional score. Each participant's outcome is compared to every other participant's outcome, assigned a score, and the summed scores are ranked. The mean rank score for each treatment group can then be calculated. A higher mean CAFS rank score indicates a better group outcome. The survival outcome is death or death-equivalent, where a participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row. The functional outcome is the ALS Functional Rating Scale-Revised (ALSFRS-R) score with a maximum total score of 48 and a minimum total score of 0. Participants with higher scores have more physical function.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Rank
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Rank | 152.10 (9.622) | 162.39 (7.328)
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.4074, Mixed Models Analysis; Covariates: baseline (BL) of use edaravone, riluzole, & Relyvrio, BL log NfL, and TRICALS score; Mean Difference (Net) = -10.29, 95% CI 2-sided [-34.69 to 14.11], Standard Error of Mean 12.401 — DNL343 24-week change from baseline relative to placebo 24-week change from baseline; Model adjusted for baseline (BL) of use edaravone, riluzole, & Relyvrio, baseline log NfL, and TRICALS score

4. Secondary Outcome: Respiratory Function
Description: Change in respiratory function over time as assessed by slow vital capacity (SVC)
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 24-week diff. of percents of normal VC
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
24-week diff. of percents of normal VC | -12.259 (1.4904) | -9.692 (1.6572)
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.2856, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -2.568, 95% CI [-7.291 to 2.156], Standard Error of Mean 2.4001 — DNL343 24-week change from baseline relative to placebo 24-week change from baseline; The model include fixed terms for regimen, visit, treatment group, treatment group × visit interaction, baseline score and baseline score x visit interaction, baseline TRICALs risk score and baseline TRICALS risk score × visit interaction, baseline riluzole use and baseline riluzole use × visit interaction, baseline edaravone use and baseline edaravone use × visit interaction, baseline Relyvrio use and baseline Relyvrio × visit interaction, and baseline log-transformed serum NfL level and baseline log-transformed serum NfL level × visit interaction

5. Secondary Outcome: Upper Limb Muscle Strength
Description: Change in upper limb muscle strength over time as measured isometrically using hand-held dynamometry and grip strength, calculated as the average percent change from baseline of the following muscles/maneuvers: shoulder flexion, elbow flexion, elbow extension, wrist extension, abductor pollicis brevis contraction, abductor digiti minimi contraction, first dorsal interosseous contraction, and grip strength. Note that only those with measurable strength at baseline were included.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Percent change | -33.787 (2.4649) | -38.573 (2.7828)
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.2318, Mixed Models Analysis; Covariates: baseline (BL) of use edaravone, riluzole, & Relyvrio, BL log NfL, and TRICALS score and interaction with visit; Mean Difference (Net) = 4.785, 95% CI 2-sided [-3.071 to 12.642], Standard Error of Mean 3.9949 — DNL343 24-week change from baseline relative to placebo 24-week change from baseline; [other analysis details as in outcome 4, analysis 1]

6. Primary Outcome: Mortality Event Rate
Description: The Mortality Rate, presented as mean deaths per month, was estimated from a Bayesian shared-parametric model that assumed exponentially distributed survival times. Mortality is defined as death or death equivalent. A participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Events per month
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Events per month | 0.007 (0.0021) | 0.007 (0.0020)

7. Secondary Outcome: Number of Participants With Death or Permanent Assisted Ventilation (PAV)
Description: The number of participants who died or met the criterion for a death equivalent from the date of their baseline visit to the end of the Week 24 visit window (generally 175 days after baseline). The death equivalent criterion is use of permanent assisted ventilation (PAV) for more than 22 hours per day for more than 7 days in a row.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Participants | 8 | 5
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.7628, Log Rank

8. Secondary Outcome: Number of Participants Who Experience Death
Description: The number of participants who died from the date of their baseline visit to the end of the Week 24 visit window (generally 175 days after baseline).
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
Participants | 6 | 4
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.8662, Log Rank

9. Secondary Outcome: Disease Progression Biomarker
Description: Change in log-transformed serum neurofilament light protein (NfL) concentration from baseline to Week 24
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | DNL343 | Matching Placebo
Number analyzed (Participants) | 186 | 139
ng/L | 0.074 (0.0224) [1.031 to 1.125] | -0.006 (0.0256) [0.945 to 1.045]
Statistical Analysis 1: Comparison: DNL343 vs Matching Placebo; Test type: Superiority; p = 0.0304, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = 0.080, 95% CI 2-sided [0.008 to 0.152]; [other analysis details as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 35 weeks after participant signed Master Protocol consent. For safety analyses, the analysis populations include all anticipated and unanticipated safety events (i.e. Deaths, Serious Adverse Events, and Other Adverse Events) due to any cause, that occurred or worsened on or after treatment initiation to either the final safety visit, the date of death, the date of last study contact, or the date of first dose of study drug during participation in the ATE period.
Description: The all-cause mortality data was analyzed using the Efficacy Regimen Only (ERO) set, which excludes placebo participants from other regimens, and includes all anticipated and unanticipated safety events that occurred within the safety analyses time frame.
Arm/Group | DNL343 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 6/186 | 3/63
Serious Adverse Events (participants affected / at risk) | 28/186 | 10/63
Other Adverse Events (participants affected / at risk) | 149/186 | 43/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DNL343 (N=186) | Matching Placebo (N=63)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug eruption (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DNL343 (N=186) | Matching Placebo (N=63)
Constipation (Gastrointestinal disorders) | 30 (31) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 20 (25) | 8 (10)
Nausea (Gastrointestinal disorders) | 17 (19) | 4 (4)
Salivary hypersecretion (Gastrointestinal disorders) | 14 (14) | 2 (2)
Fatigue (General disorders) | 41 (49) | 10 (10)
COVID-19 (Infections and infestations) | 14 (14) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (14) | 3 (7)
Urinary tract infection (Infections and infestations) | 19 (23) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 73 (154) | 13 (17)
Cognitive disorder (Nervous system disorders) | 11 (11) | 1 (1)
Dizziness (Nervous system disorders) | 14 (16) | 1 (1)
Headache (Nervous system disorders) | 30 (36) | 10 (16)
Muscle contractions involuntary (Nervous system disorders) | 10 (10) | 5 (5)
Muscular weakness (Nervous system disorders) | 42 (82) | 6 (13)
Neuromyopathy (Nervous system disorders) | 11 (12) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 12 (12) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (5)
Anxiety (Psychiatric disorders) | 10 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05842941/Prot_002.pdf
  • Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT05842941/SAP_001.pdf